CLINICAL TRIAL: NCT02595125
Title: Comparative Study, Prospective, Randomized , Assessing the Reduction of Pain Felt During Installation Intra- Uterine Device by Direct Technique. A Monocentric Study
Brief Title: Study Assessing the Reduction of Pain Felt During Installation Intra- Uterine Device by Direct Technique
Acronym: DIRECTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1508153; 2015-A01966-43 (Other: ANSM)
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Contraception
Keywords: intrauterine device; contraceptive method; direct technique; torpedo technique; verbal numeric scale

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional technique (Sham Comparator): Intrauterine device (IUD) insertion by the conventional technique
  Interventions: Device: IUD
- Direct technique (Experimental): Intrauterine device (IUD) insertion by the direct technique
  Interventions: Device: IUD

INTERVENTIONS:
Device: IUD — copper IUD or levonogestrel IUD insert by the conventional technique or by direct technique

SUMMARY:
Intrauterine devices (IUDs) are contraceptive methods of long-acting (from 3 to 10 years depending on the model) and among the most effective. However, there are many obstacles to the use of IUDs including pain felt by patients during installation. Several medical means were studied without evidence of their efficacy in pain related to IUD insertion. In order to remove this brake, it's important to find another way to act against this pain. The direct technique is one of the techniques described by health professionals. It seems trusted by its users as a more reliable technique but also less painful for patients. However, there is no study available on its evaluation. The aim of this study is to investigate the interest of the direct technique in reducing the pain experienced by patients during installation.

ELIGIBILITY:
Inclusion Criteria:

* Any major patient and consultant for IUD insertion : hormonal or copper
* Signing of the information and consent form by the patient or, if under supervision by parents or guardian.
* Patient affiliated with or entitled to a social security scheme
* No contraindication for IUD insertion

Exclusion Criteria:

* Patient consultant for IUD insertion to side arms
* Contraindications for installation.
* Legal incapacity or limited legal capacity. Medical or psychological conditions not allowing the subject to understand the study and sign the consent
* Refusal to sign the consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Pain measured by Verbal Numeric Scale | intraoperative
  Pain is score by Verbal Numeric Scale : 0-10 (0 = no pain; 10= pain as bad as can be)

SECONDARY OUTCOMES:
Number of failure laying direct technique | intraoperative
Number of vagal discomfort | intraoperative
Number of expulsion of the IUD | intraoperative
Number of IUD-fond uterine distance >2 cm | intraoperative
Number of expulsion of IUD | up to 7 days
Number of emergency department visit for a IUD complication | up to 7 days
Number of analgesic intake | up to 7 days post-insertion
Pain measured by Verbal Numeric Scale | day 1
  Pain is score by Verbal Numeric Scale : 0-10 (0 = no pain; 10= pain as bad as can be)
Pain measured by Verbal Numeric Scale | day 7
  Pain is score by Verbal Numeric Scale : 0-10 (0 = no pain; 10= pain as bad as can be)

CONTACTS AND LOCATIONS:
Overall Officials: Céline Chauleur, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No